CLINICAL TRIAL: NCT03571126
Title: Olanzapine as First Line Treatment for Prevention of Nausea and Vomiting Induced by Chemotherapy of Lung Cancer: a Multicenter, Double-blind and Randomized Trial
Brief Title: Olanzapine for the Prevention and Treatment of Nausea and Vomiting Induced by Chemotherapy of Lung Cancer
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zunyi Medical College (Other)
Collaborators: Zunyi First People's Hospital (Industry); Afﬁliated Hospital of North Sichuan Medical College (Other); Sichuan Cancer Hospital and Research Institute (Other); Guizhou Provincial People's Hospital (Other); Affiliated Hospital of Southwest Medical University (Other)
Responsible Party: Principal Investigator, Jian-Guo Zhou,MD, Principal Investigator, Zunyi Medical College
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 20180520
Record Dates: First submitted 2018-06-07; First posted 2018-06-27 (Actual); Last update posted 2021-07-13 (Actual); Status verified 2021-07

CONDITIONS: Chemotherapy-induced Nausea and Vomiting; Lung Cancer
MeSH Terms: conditions — Vomiting; Lung Neoplasms | interventions — Olanzapine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebos group (Placebo Comparator): Patients will be administered with dexamethasone plus tropisetron from D1 to D3.
  Patients will also be administrated with placebos from D1-D4
  Interventions: Drug: Placebos
- Experimental group (Experimental): Patients will receive a regimen with dexamethasone plus tropisetron from D1-D3. Patients will also be administrated with olanzapine from D1-D4.
  Interventions: Drug: Olanzapine

INTERVENTIONS:
Drug: Olanzapine — Dexamethasone (10mg/d) (Days1-3) Tropisetron (4mg or 4.48mg or 5mg /d) (Days1-3) Olanzapine (10mg/d) (Days1-4)
  Arms: Experimental group
Drug: Placebos — Dexamethasone (10mg/d) (Days1-3) Tropisetron (4mg or 4.48mg or 5mg /d) (Days1-3) Placebos (Days1-4)
  Arms: Placebos group

SUMMARY:
Chemotherapy induced nausea and vomiting (CINV) is a common adverse effect in treatment of cancer, which influences the quality of life and adherence to treatment of patients and leads to dehydration, malnutrition and even death. Prevention and relieving the CINV is an important step to ensure the conduction of chemotherapy. Mechanism of CINV remains to be obscure, while most studies showed that it is mainly related to the following respects: ⑴ Chemotherapeutic agents stimulate gastrointestinal tract, which induces the release of neurotransmitters by chromaffin cells. Neurotransmitters bind to corresponding receptors, and then results in vomiting by stimulating the vomiting center; ⑵ Chemotherapeutic agents and the metabolites of them activate chemoreceptors directly, which causes vomiting. ⑶ Feeling and mental factors irritate cerebral cortex pathway directly. There are studies suggested that 5- hydroxytryptamine (5-HT) was related to acute nausea and vomiting induced by chemotherapy, which means 5-HT receptor antagonist would be a effective medicine for acute CINV. In addition, there are researches proclaimed that neurokinin-1 (NK-1) receptor antagonist, aprepitant, is a potent agent to relieve CINV. Thus, correlative guidelines recommend regimens with 5-HT receptor antagonist, NK-1 receptor antagonist and glucocorticoid as the standard treatment for strongly emetic chemotherapy regimens. But the prevention of moderately emetic chemotherapy regimens remains to be a problem in clinical practice. Besides, there is no study to demonstrate differences of mechanisms between acute CINV and delayed CINV. Olanzapine inhibits kinds of neurotransmitters which cause CINV, it is why this medicine is effective in both acute and delayed CINV. It can also alleviate anxiety, improve sleep quality and relieve pain in patients with cancer. The most common adverse effects of olanzapine are lethargy, body mass increase, fatigue, dry mouth, constipation, hyperlipidemia and hyperglycemia. Among them, the most common one is lethargy, which can oppose insomnia and excitation caused by dexamethasone. In a word, olanzapine is an agent with mild adverse effects, it is worth to be generalized. But there are still problems to be resolved in the application of olanzapine in CINV: ⑴ Aprepitant is expensive and not covered in medical care in China, which limits the application in patients. ⑵There is no large clinical trial to confirm the efficacy and safety of olanzapine in Chinese populations. To explore these issues better, investigators intend to compare the regimen with olanzapine, dexamethasone and 5-HT receptor antagonists with the regimen with placebo, dexamethasone and 5-HT receptor antagonists about the efficacy and adverse events in treatment of CINV. Investigators aim to provide an available therapeutic options for CINV, improve the quality of life and prolong the survival of patients with lung cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Eastern Cooperative Oncology Group (ECOG) Performance Status≤2 or Karnofsky performance statu (KPS) scores≥60.
2. Patients with cytologically or histologically confirmed lung cancer.
3. Patients who are willing to receive chemotherapy and can tolerate at least 2 cycles chemotherapy.
4. Chemotherapy regimens accord with standard regimens recommended by clinical practice guidelines (National Comprehensive Cancer Network guidelines and Chinese Society of Clinical Oncology guidelines of lung cancer).
5. There is at least one kind of high emetic risk chemotherapy agent, mainly including regimens contain cisplatin or carboplatin (AUC≥4).
6. Adequate organ function including the following: Adequate bone marrow reserve: white blood cell (WBC) count superior or equal to 2.0×10^9/L , absolute neutrophil count (ANC) superior or equal to 1.5×10^9/L, platelets superior or equal to 80×10^9/L, and hemoglobin superior or equal to 90g/L; Hepatic: bilirubin <1.5 times the upper limit of normal (ULN), aspartate transaminase (AST) and alanine transaminase (ALT) ≤2.5×ULN (or <5×ULN with liver metastases); Renal: Serum creatinine≤1×ULN, calculated creatinine clearance (CrCl) superior or equal to 50 milliliter/min based on the standard Cockcroft and Gault formula.
7. At least 3 weeks after the end of the last chemotherapy.
8. Women of reproductive years are willing to contracept in appropriate methods in the period of trial and in the 8 weeks after the last administration. Doing pregnancy test before the beginning of this trial when necessary, and results of which need to be negative.

Exclusion Criteria:

1. Women who are pregnant or breastfeeding
2. Need to undergo radiotherapy during this trial.
3. Patients with alimentary tract obstruction.
4. Patients with severe heart disease, renal and liver disease and metabolic abnormalities.
5. Patients with epilepsy or who are using antipsychotics.
6. Patients who have been administrated with antiemetic in 24 hours or who have suffered vomiting before chemotherapy.
7. Patients with brain metastases.
8. Patients with contraindications of chemotherapy.
9. Patients who are attending another clinical trial or will attend in 2 weeks.
10. Patients who are considered unsuitable to be included by treating physicians.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 156 (Estimated)
Dates: Start 2019-05-09 (Actual); Primary Completion 2022-10-01 (Estimated); Study Completion 2023-08-01 (Estimated)

PRIMARY OUTCOMES:
Incidence rate of no delayed nausea and vomiting | 1 week
  Number of participants with nausea and vomiting occuring within 24 hours after chemotherapy in all participants.

SECONDARY OUTCOMES:
Complete response of acute nausea and vomiting | 1 week
  Number of participants with no nausea and vomiting occuring within 24 hours after chemotherapy as assessed by CTCAE v4.0.
Complete response of delayed nausea and vomiting | 1 week
  Number of participants with no nausea and vomiting occuring in 24 hours to 120 hours after chemotherapy as assessed by CTCAE v4.0.
Disease control rate | 1 week
  Number of participants who reach complete response or partial response.
Quality of life of participants by The European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire-Lung Cancer 13 scale | 1 week
  Quality of life of participants is measured with The European Organisation for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire-Lung Cancer 13(QLQ-LC13) scale which is filled by participants themselves. The questionnaire is consist of several symptoms measured by scores range from 1 to 7, the higher the symptoms are scored, the worse the quality of life is.
Quality of life of participants by The European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire-Lung Cancer 30 scale | 1 week
  Quality of life of participants is measured with EORTC QLQ-LC30 scale which is filled by participants themselves. The questionnaire is consist of several symptoms measured by scores range from 1 to 7, the higher the symptoms are scored, the worse the quality of life is.
Quality of life of participants by Functional Assessment of Cancer Therapy-Lung cancer scale | 1 weeks
  Quality of life of participants is measured with Functional Assessment of Cancer Therapy-Lung cancer (FACT-L) scale which is filled by participants themselves. The FACT-L, version 4, is a combination of the 27-item FACT-General (FACT-G) and the 9-item Lung Cancer Subscale (LCS) which measures multidimensional quality of life. The FACT-L score ranges from 0 to 136. The higher the score obtained by each patient in question, the greater the final score of the subscale and the better the quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Hu Ma, Doctor, Principal Investigator — Zunyi Medical College
Locations (2):
- China (2):
  - Affiliated Hospital of Zunyi Medical University, Zunyi, Guizhou
  - Afﬁliated Hospital of North Sichuan Medical College, Nanchong, Sichuan

IPD SHARING:
Plan to Share IPD: Yes
The individual participant data will be available to other researchers in this study and physicians treating study participants.Jiangsu Famous Medicine Co.,Ltd. provide EDC.
Supporting Information: Study Protocol, ICF, CSR
Time Frame: 5 months after publication.
Access Criteria: the physician treating the study participants and other researchers in this study will receive a report that summarizes the findings of this study.

REFERENCES:
- [Background] Hesketh PJ, Kris MG, Basch E, Bohlke K, Barbour SY, Clark-Snow RA, Danso MA, Dennis K, Dupuis LL, Dusetzina SB, Eng C, Feyer PC, Jordan K, Noonan K, Sparacio D, Somerfield MR, Lyman GH. Antiemetics: American Society of Clinical Oncology Clinical Practice Guideline Update. J Clin Oncol. 2017 Oct 1;35(28):3240-3261. doi: 10.1200/JCO.2017.74.4789. Epub 2017 Jul 31. PMID 28759346
- [Background] Adel N. Overview of chemotherapy-induced nausea and vomiting and evidence-based therapies. Am J Manag Care. 2017 Sep;23(14 Suppl):S259-S265. PMID 28978206
- [Background] Navari RM. 5-HT3 receptors as important mediators of nausea and vomiting due to chemotherapy. Biochim Biophys Acta. 2015 Oct;1848(10 Pt B):2738-46. doi: 10.1016/j.bbamem.2015.03.020. Epub 2015 Mar 30. PMID 25838122
- [Background] Navari RM, Gray SE, Kerr AC. Olanzapine versus aprepitant for the prevention of chemotherapy-induced nausea and vomiting: a randomized phase III trial. J Support Oncol. 2011 Sep-Oct;9(5):188-95. doi: 10.1016/j.suponc.2011.05.002. Epub 2011 Sep 24. PMID 22024310
- [Background] Geling O, Eichler HG. Should 5-hydroxytryptamine-3 receptor antagonists be administered beyond 24 hours after chemotherapy to prevent delayed emesis? Systematic re-evaluation of clinical evidence and drug cost implications. J Clin Oncol. 2005 Feb 20;23(6):1289-94. doi: 10.1200/JCO.2005.04.022. PMID 15718327
- [Background] Walsh D, Davis M, Ripamonti C, Bruera E, Davies A, Molassiotis A. 2016 Updated MASCC/ESMO consensus recommendations: Management of nausea and vomiting in advanced cancer. Support Care Cancer. 2017 Jan;25(1):333-340. doi: 10.1007/s00520-016-3371-3. Epub 2016 Aug 17. PMID 27534961
- [Background] Passik SD, Kirsh KL, Theobald DE, Dickerson P, Trowbridge R, Gray D, Beaver M, Comparet J, Brown J. A retrospective chart review of the use of olanzapine for the prevention of delayed emesis in cancer patients. J Pain Symptom Manage. 2003 May;25(5):485-8. doi: 10.1016/s0885-3924(03)00078-2. PMID 12727048
- [Background] Zhang Z, Zhang Y, Chen G, Hong S, Yang Y, Fang W, Luo F, Chen X, Ma Y, Zhao Y, Zhan J, Xue C, Hou X, Zhou T, Ma S, Gao F, Huang Y, Chen L, Zhou N, Zhao H, Zhang L. Olanzapine-Based Triple Regimens Versus Neurokinin-1 Receptor Antagonist-Based Triple Regimens in Preventing Chemotherapy-Induced Nausea and Vomiting Associated with Highly Emetogenic Chemotherapy: A Network Meta-Analysis. Oncologist. 2018 May;23(5):603-616. doi: 10.1634/theoncologist.2017-0378. Epub 2018 Jan 12. PMID 29330211